CLINICAL TRIAL: NCT07198828
Title: Development and Evaluation of a Mobile Health (mHealth) Application for Smoking Cessation Among Adolescents in Indonesia: A Mixed Methods Randomized Controlled Trial
Brief Title: Mobile Health (mHealth) Application for Smoking Cessation Among Adolescents in Indonesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Radian Ilmaskal, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KE-FK-0864-EC-2025
Record Dates: First submitted 2025-09-16; First posted 2025-09-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Tobacco Use Disorder; Smoking Cessation; Adolescent Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth Intervention Group (Experimental): Participants receive the mHealth smoking cessation application with:
  * Educational content about smoking risks and cessation benefits
  * Motivational messages and progress tracking
  * Social support features
  * Interactive elements and quizzes
  * Monthly monitoring and support
  Interventions: Behavioral: mHealth Smoking Cessation Application
- Control Group (Active Comparator): Participants receive paper-based smoking cessation module containing equivalent content:
  * Motivational content and cessation benefits
  * Ex-smoker success stories
  * Trigger identification and coping strategies
  * Weekly quizzes with prizes (online access)
  * Monthly check-ins
  Interventions: Behavioral: Paper-based Control Materials

INTERVENTIONS:
Behavioral: mHealth Smoking Cessation Application — Participants receive the mHealth smoking cessation application with:
  * Educational content about smoking risks and cessation benefits
  * Motivational messages and progress tracking
  * Social support features
  * Interactive elements and quizzes
  * Monthly monitoring and support
  Arms: mHealth Intervention Group
Behavioral: Paper-based Control Materials — Participants receive paper-based smoking cessation module containing equivalent content:
  * Motivational content and cessation benefits
  * Ex-smoker success stories
  * Trigger identification and coping strategies
  * Weekly quizzes with prizes (online access)
  * Monthly check-ins
  Arms: Control Group

SUMMARY:
This mixed-methods study develops and evaluates a mobile health (mHealth) application for smoking cessation among Indonesian adolescents aged 13-15 years. The study uses a sequential exploratory approach with three phases: (1) qualitative research to inform app design; (2) app development using Rapid Application Development (RAD) model; and (3) a single-blind, two-arm randomized controlled trial comparing the mHealth intervention to paper-based materials. The intervention is grounded in the Unified Theory of Acceptance and Use of Technology (UTAUT2) and Transtheoretical Model (TTM). Primary outcome is smoking abstinence at 1-, 3-, and 6-month follow-ups measured through self-report questionnaires.

DETAILED DESCRIPTION:
Adolescent smoking is a growing public health concern worldwide, and it is particularly prevalent in low- and middle-income countries (LMICs) such as Indonesia. According to the World Health Organization (WHO), nearly 6.5% of adolescents aged 13-15 years globally use tobacco, with Southeast Asia, including Indonesia, contributing a significant proportion of this population. The prevalence of smoking among Indonesian adolescents has escalated over the past decade, with national surveys indicating a sharp increase from 7.2% in 2013 to 9.1% in 2018 and even higher figures reported by the 2019 Global Youth Tobacco Survey (GYTS) at 19.2%. Although more recent estimates suggest a slight reduction to 7.4% in 2023, smoking among adolescents remains a major public health challenge in Indonesia. Especially since Indonesia is the only country in Asia that has not ratified the WHO Framework Convention on Tobacco Control (FCTC).

This condition is especially concerning given the strong empirical evidence of the detrimental effects of smoking on individual health, societal well-being, and the environment. Adolescent smoking is associated with numerous long-term health risks, including respiratory diseases, cardiovascular problems, and an increased likelihood of continuing smoking into adulthood. Furthermore, smoking during adolescence has been linked to mental health issues such as depression, anxiety, and suicidal ideation. Moreover, tobacco-related mortality is alarmingly high, with over 8 million deaths annually worldwide due to active smoking and exposure to secondhand smoke. In Indonesia, tobacco-related diseases contribute significantly to mortality, with an estimated 225,700 deaths annually attributed to smoking. Despite various tobacco control measures implemented in Indonesia, such as raising taxes on tobacco products, free smoking cessation consultation services, and establishing smoke-free zones, smoking rates among adolescents have remained persistently high.

Technology-based interventions, particularly mobile health (mHealth) applications, have emerged as promising tools for promoting smoking cessation. The widespread use of smartphones among adolescents, with Indonesia being the fourth-largest smartphone market globally, presents a unique opportunity to leverage mHealth interventions to reduce smoking rates. However, the effectiveness of mHealth applications for smoking cessation has shown inconsistent results, particularly in LMICs where accessibility, engagement, and content relevance may differ from those in high-income countries.

Previous studies have demonstrated that while mHealth applications can help individuals quit smoking in the short term, their long-term effectiveness remains unclear, especially among adolescent populations. There is a growing body of literature highlighting the importance of tailoring interventions to the unique needs of adolescents, taking into account developmental stages, peer influence, and social media dynamics. However, there is a significant gap in the availability of mHealth applications designed specifically for adolescents in Indonesia, and the existing tools often fail to integrate critical elements such as behavioral change techniques, social support, and interactive features.

This study aims to address these gaps by developing an innovative mHealth intervention designed specifically for adolescent smokers in Indonesia. The intervention will be grounded in behavioral change theories such as the Unified Theory of Acceptance and Use of Technology (UTAUT2) and the Transtheoretical Model (TTM). UTAUT2 will ensure that the app is accepted, used, and engaging for adolescents, taking into account the influence of peers, ease of use, and intrinsic motivation factors. TTM will guide the app design by allowing it to adapt to the adolescent's specific stage in the smoking cessation process, providing tailored content and support. Together, these frameworks will make the mHealth app both effective, promoting long-term behavior change, relevant for adolescent smokers and better smoking cessation outcomes in Indonesia.

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1 (Qualitative Study):

   * Adolescent smokers aged 13-15 years
   * Smoking at least one cigarette or vaping once per week
   * Key informants: teachers, parents, peers, healthcare workers with relevant experience
2. Phase 3 (RCT):

   * Adolescents aged 13-15 years
   * Smoking at least 1 cigarette in the past week
   * Own smartphone with internet access
   * Living in Padang City during study period
   * Willing to participate until study completion
   * Desire to quit smoking

Exclusion Criteria:

Phase 3 (RCT):

* Currently using other smoking cessation apps or programs
* Planning to change schools or relocate outside Padang during study period
* Have severe psychiatric or medical conditions requiring intensive treatment
* Unable to use smartphone applications due to literacy or technical limitations

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported smoking abstinence measured through questionnaire (Yes/No response where Yes = abstinent, No = not abstinent) | 1, 3, and 6 months post-intervention

SECONDARY OUTCOMES:
Smoking cessation self-efficacy using SEQ-12 (12-item Smoking Self-Efficacy Questionnaire) | Baseline, 1, 2, 3, and 6 months
  Scale range: 12-60, where higher scores indicate greater self-efficacy for smoking cessation
Motivation assessed via Richmond Test | Baseline, 1, 2, 3, and 6 months
  Scale range: 0-10, where higher scores indicate greater motivation to quit smoking
Social support measured through Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline, 1, 2, 3, and 6 months
  Scale range: 12-84, where higher scores indicate greater perceived social support
Dependence level using Fagerström Test for Nicotine Dependence (FTND) | Baseline, 1, 2, 3, and 6 months
  Scale range: 0-10, where higher scores indicate greater nicotine dependence
App usage engagement measured through usage logs | Baseline, 1, 2, 3, and 6 months
  Frequency and duration of app usage tracked through automated logging system. Measured as number of sessions per week and average session duration in minutes
mHealth app usability measured through mHealth Usability Questionnaire (MAUQ) | Time Frame: 1, 2, 3, and 6 months
  mHealth Usability Questionnaire (MAUQ) scores. Scale range: 18-126, where higher scores indicate better perceived usability of the mobile health application

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple junior high schools and community health centers, Padang, West Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie the results reported in this article, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to yayisuryo@ugm.ac.id. Data requestors will need to sign a data access agreement.